CLINICAL TRIAL: NCT04645914
Title: Laser Speckle Contrast Analysis to Evaluate the Influence of the Consumption of Conventional and Electric Cigarettes on Skin Circulation
Brief Title: Influence of the Consumption of Conventional and Electric Cigarettes on Skin Circulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Andreas Kyriakou, Vacular Surgery Resident, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Laser Doppler Camera Study 1
Record Dates: First submitted 2020-11-15; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Nicotine Dependence; Vaping; Smoking
Keywords: Perfusion; Laser Speckle Contrast Analysis; Laser Doppler Camera; Nicotine; Smoking; Vaping
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Smoking | interventions — Smoking Devices; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Two groups : consumers of cigarettes/e-cigarettes and non consumers of cigarettes/e-cigarettes
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind through randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No smokers (No Intervention): Healthy subjects who do not consume any nicotine products
- Smokers/Vapers (Experimental): Healthy subjects who consume nicotine products
  Interventions: Behavioral: Use of nicotine product (smoking/vaping)

INTERVENTIONS:
Behavioral: Use of nicotine product (smoking/vaping) — The smokers/vapers are consuming during the study one nicotine product of their own. The dose is the same as each individual is consuming regularly
  Arms: Smokers/Vapers

SUMMARY:
The survey participants are divided into a smoking and non-smoking group. The smoker group is further divided according to the quantity and quality of nicotine ("normal" smoking, vaping). After reaching a steady state, the cutaneous blood flow at rest in the extremities of all participants is determined by Laser Doppler Imaging as a reference value. Laser Doppler Imaging produces images of the blood flow using perfusion units (PU). Subsequently, the perfusion is measured again after smoking/vaping. The difference in skin perfusion of the extremities is calculated (δ-Perfusion). All measurements are performed under controlled vital parameters (body temperature, systolic and diastolic blood pressure, heart rate) and controlled room temperature as well as 15-minute acclimatization of the patients.

DETAILED DESCRIPTION:
After consenting to the study, the subjects are examined using Laser Doppler Camera.

The skin blood flow of the extremities is determined as a reference value. Laser Doppler Imaging produces images of the blood flow using the perfusion units (PU).

All measurements are taken under controlled vital parameters (body temperature, systolic and diastolic blood pressure, heart rate) and controlled room temperature as well as 15-minute acclimatization of the subjects.

For smokers or vapers, the perfusion is measured again after consuming a cigarette or an e-cigarette respectively. The difference of blood flow after smoking or vaping is calculated using both measures.

The total duration of the study per subject is approximately 25-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult non-smokers, smokers, vapers

Exclusion Criteria:

* Adults with cardiopulmonary diseases
* Pregnant women
* Adults that participating in other surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Perfusion of the extremities for non-smokers, smokers and vapers | 30 seconds
  The perfusion of the extremities will be measured in Perfusion Units. The Perfusion Units are calculated directly through the Laser Doppler Camera as a result of the examination.
Difference of perfusion after smoking/vaping | 30 seconds
  The perfusion of the extremities will be measured after the consume of cigarettes/electronic cigarettes in Perfusion Units. The difference between the results of the examination before and after the consume of cigarettes/electronic cigarettes will be measured in Perfusion Units.

SECONDARY OUTCOMES:
Correlation of perfusion with age | 30 seconds
  The age (years) will be controlled as a possible factor that influence the perfusion. Therefore the results in Perfusion Units measured through Laser Doppler Camera will be statistically analyzed taking into consideration the age in years of each subject.
Correlation of perfusion with gender | 30 seconds
  The gender(male or female) will be controlled as a possible factor that influence the perfusion. Therefore the results in Perfusion Units measured through Laser Doppler Camera will be statistically analyzed taking into consideration the gender of each subject.
Correlation of perfusion with quantity of smoking/vaping | 30 seconds
  The quantity of smoking/vaping (packet years/nicotine quantity for vaping) will be controlled as apossible factor that influence the perfusion. Therefore the results in Perfusion Units measured through Laser Doppler Camera will be statistically analyzed taking into consideration the quantity of smoking of each related subject.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kyriakou, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No